CLINICAL TRIAL: NCT01066832
Title: The Valentines Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eurocor GmbH (Industry)
Responsible Party: Dr. Rembert Pogge von Strandmann, Eurocor GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eur-001
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2010-02

CONDITIONS: Instent Restenosis
Keywords: Drug-eluting balloon; Paclitaxel; DIOR; short term registry; Valentines Trial; Drug-eluting balloon treatment of in-stent restenosis
MeSH Terms: interventions — Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel-coated balloon (3 µg/mm2)

SUMMARY:
The primary objective of this multi-center, international, short term registry is to assess clinical success and efficacy of the paclitaxel eluting balloon treatment for in-stent restenosis at 6-9 months follow up. Clinical success defined as freedom from major adverse cardiac events (MACE: death, myocardial infarction [MI], target lesion revascularization [TLR]) and target vessel revascularization [TVR]) and stent thrombosis, both early and late occurrences will be assessed.

In addition, a cohort of the registry will undergo angiographic follow up at 6-9 months to assess in-stent and in-segment late loss and binary restenosis subsequent to paclitaxel eluting balloon treatment for in-stent restenosis.

A prioi analysis will be comparison of the safety and efficacy of patients presenting with drug-eluting stent in-stent restenosis to bare metal stent in-stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, > 18 years of age;
* Patients who present with in-stent restenosis of a previously placed stent documented by coronary angiogram for which re-PCI is planned;
* The patient has stable or unstable angina, and/or clinical evidence of ischemia (ECG, exercise test, etc.);
* The target lesion is in a native vessel;
* Up to two lesions per patient;
* Target lesion(s) stenosis is > 50%.

Exclusion Criteria:

* The patient has had an acute myocardial infarction within the last 48 hours;
* The patient has a co-morbid illness (i.e. any illness likely to limit his/her life expectancy to <12 months);
* Lesion(s) requiring additional stenting either bare metal or drug eluting (non, bail-out indications);
* The patient has had previous therapeutic radiation to the target vessel;
* The patient is unable the take dual antiplatelet therapy for at least 6 months;
* Patients with three or more lesions with in-stent restenosis requiring angioplasty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Clinical success at 6-9 month defined as freedom from MACE, death, MI,TLR and stent thrombosis | 6-9 month

SECONDARY OUTCOMES:
In-stent and in-segment late loss and binary restenosis | 6-9 month

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Stella, MD, PhD, Principal Investigator — UMC Utrecht, Utrecht, Netherlands; Sigmund Silber, Prof., Principal Investigator — Heart Center Munich at the Isar, Munich, Germany; Giuseppe Sangiorgi, MD, Principal Investigator — Policlinico Modena, Modena, Italy
Locations (3):
- Heart Center Munich at the Isar, Munich, Germany
- Policlinico, Modena, Italy
- UMC Utrecht, Utrecht, Netherlands